CLINICAL TRIAL: NCT03808168
Title: Phase II Trial of Nivolumab Based Immunotherapy for the Treatment of High-Grade Cervical Dysplasia
Brief Title: Nivolumab Based Immunotherapy for Treatment of High Grade Cervical Dysplasia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA has withdrawn the IND application- requesting protocol changes
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 032017-028
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Cervix Uteri--Diseases
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Nivolumab, 3 mg/kg Iv, day 1
  Interventions: Drug: Nivolumab
- Arm 2 (Active Comparator): Nivolumab, 3 mg/kg IV, days 1, 15, 29
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Protocol dose: 3mg/kg mg as a 30-minute IV infusion on Day 1 (Arm I) or Days 1, 15, 29 (Arm II).
  Other Names: Opdivo, BMS-936558, MDX1106

SUMMARY:
The study design is a phase II interventional trial for women with biopsy proven high-grade cervical dysplasia. The study is an open label study and randomized. The study will have two arms. Patients will be randomized to both arms.

DETAILED DESCRIPTION:
High-grade cervical dysplasia (cervical intraepithelial neoplasia (CIN) II/III), is both detectable and quantifiable, which presents many opportunities for evaluation or early treatment, intervention and eventually, for cancer prevention. High-grade dysplasia is typically detected during cervical cancer screening with a pap smear. To determine the pathologic response rate of high grade cervical dysplasia with PD-1 checkpoint modulation with Nivolumab.This is a randomized phase II trial with two experimental arms (1 dose of nivolumab and 3 doses of nivolumab).

ELIGIBILITY:
Inclusion Criteria:

* Adult female subjects (age 18 years or older)
* Performance status ECOG 0-1
* All patients must have cervical biopsies demonstrating high-grade cervical dysplasia.
* All patients must have a satisfactory colposcopy with visualization of the entire squamo-columnar junction
* All patients must be candidates for a cervical conization procedure or LEEP procedure
* The patient is able and willing to comply with study procedures, and signed and dated informed consent is obtained before any study-related procedure is performed
* Negative screening test results for hepatitis B, hepatitis C, and human immunodeficiency virus
* At least six weeks must have elapsed from any prior chemotherapy, radiation therapy or immunotherapy
* Patients must have adequate:

  * Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl. Platelets greater than or equal to100, 000/mcl. Hemoglobin > 9 gm/dL.
  * Renal function: creatinine less than or equal to institutional upper limit normal (ULN) or calculated creatinine clearance (Cockcroft-Gault) ≥ 50 ml/min.
  * Serum creatinine </= 1.5xULN or creatinine clearance (CrCl) >/=50 mL/min (using the Cockcroft-Gault formula)
  * Female CrCl = (140-age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Metabolic function: Calcium, Magnesium, Phosphate, and Potassium levels within institutional normal limits.
  * Hepatic function: Bilirubin less than or equal to 1.5 x ULN. AST and ALT less than or equal to 3 ULN and alkaline phosphatase less than or equal to 2.5 x ULN.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception. The effects of Nivolumab on the developing human fetus are unknown. For this reason and because other therapeutic agents or modalities used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, through the duration of study participation and for a period of 5 months after the last dose of nivolumab. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* The patient is lactating or pregnant
* The colposcopy is inadequate; the entire transformation zone is not visualized and endocervical curettage is positive for high-grade dysplasia
* Clinical concern for invasive cervical cancer
* Patients must not have received any prior oncology vaccine therapy
* Intercurrent medical illnesses that would impair patient tolerance to participation
* Any concurrent medical condition requiring the use of systemic steroids is not permitted (the use of inhaled or topic steroids is permitted)
* Concurrent treatment with chemotherapy, radiation therapy or immunotherapy for intercurrent illnesses
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results;
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways;
* Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll;
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Subjects with history of life-threatening toxicity, including hypersensitivity reaction, related to prior immunoglobulin treatment for another condition or any other study drug component.
* History or evidence upon physical/neurological examination of other central nervous system condition (e.g., seizures, abscess) unrelated to cancer, unless adequately controlled by medication or considered not potentially interfering with protocol treatment;
* Surgical procedure <7 days prior to study treatment, vascular access device no restriction;
* Subjects unable (e.g., due to pacemaker or ICD device) or unwilling to have a contrast-enhanced MRI of the head;
* History of allergy or hypersensitivity to study drug components
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of regression on high grade dysplasia lesions | 15 weeks after the beginning of immunotherapy
  The endpoints of the current study will be to determine the rate of spontaneous regression on high grade dysplasia lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jayanthi Lea, MD, Principal Investigator — Univeristy of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No